CLINICAL TRIAL: NCT07282639
Title: Development and Evaluation of App-Based Certified Diabetes Education (AB-CDE) Therapy for People Living With T1D Using MDI
Brief Title: App-Based Certified Diabetes Education Therapy (AB-CDE)
Acronym: AB-CDE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Leona M. & Harry B. Helmsley Charitable Trust (Unknown)
Responsible Party: Principal Investigator, Leah Wilson, Associate Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25791; 2207 (Other Grant/Funding Number: Helmsley Charitable Trust)
Record Dates: First submitted 2025-12-05; First posted 2025-12-15 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes (T1D)
Keywords: AB-CDE; DailyDose
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Intervention Group (Experimental): AB-CDE intervention using DailyDose, study CGM, and CDE and BH counselling if indicated
  Interventions: Device: DailyDose
- Control Group (No Intervention): Usual care including MDI insulin therapy with study CGM and DailyDose in Data-logging Mode.

INTERVENTIONS:
Device: DailyDose — Our team has developed a smartphone-based application, DailyDose Decision Support Tool (DailyDose), that combines continuous glucose monitoring data and insulin data to provide decision support for people living with T1D taking MDI. DailyDose is an iPhone application that is designed to support this population by 1) allowing for bolus calculation based on inputs including carbohydrate intake, CGM value and trend, and exercise information, 2) providing recommendations for carbohydrate intake based on exercise type, intensity, and duration, and 3) providing weekly recommendations for adjustments in insulin doses at specific times of day, including basal insulin dose, carbohydrate ratios or fixed mealtime doses, and correction factors .
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to learn more about a smartphone application (app) called DailyDose, an investigational decision support tool that may help in managing your diabetes. DailyDose tracks your continuous glucose monitoring (CGM) data, insulin use, and exercise, and uses this information to provide personalized recommendations for insulin dosing and carbohydrate intake during exercise or low blood sugar events. We want to find out if DailyDose can help lower blood sugar levels as measured by the hemoglobin A1c (HbA1c) test.

DETAILED DESCRIPTION:
Participants will be on study for 38 weeks (2-week run-in period and 36 weeks of intervention/control). Participants will begin the study with a training visit on the Dexcom G6 CGM system, the insulin dose capture system, and the Data-logging Mode of DailyDose. Participants will be provided with Humalog and Basaglar Tempo pens for use with the insulin dose capture system. Participants will also receive an iPhone and Apple smart watch for acquiring sleep metrics and exercise data. Participants will use these devices during the next 14 days at home (2-week run-in). At the end of the run-in, participants will be randomized to the intervention or control group. The intervention group will be trained at Visit 3 on using the DailyDose system. Participants will then use the DailyDose system for 12 weeks. Sensor glucose, exercise, insulin and meal data will be collected during the DailyDose portion of the study in order to produce recommendations for insulin dosing. Participants will wear the Dexcom G6 for the entire study. Insulin data will be collected using the insulin dose capture system (Tempo pens and Tempo button). Participants will be instructed to use the bolus calculator within the DailyDose app. Participants will be asked to complete a 30-minute aerobic exercise video at home once per week starting with the first 12-week period. After 12 weeks, time in range (70-180 mg/dL, TIR) and time in hypoglycemia (<70 mg/dL) will be assessed from the prior 4 weeks based on the Dexcom G6. Participants that have TIR ≥ 60% and time in hypoglycemia <4% will continue with use of DailyDose. Those that have TIR < 60% and/or time in hypoglycemia ≥ 4% will receive DSMES and, if recommended, behavioral health based on the T1-Diabetes Distress Assessment System (T1-DDAS) for the next 12 weeks. Additionally, if the DSMES provider feels the participant would benefit from behavioral health intervention, they can refer the participant for this even if T1-DDAS scores do not meet the cut off. All participants will then be followed for a final 12-week period using DailyDose alone to assess sustainability of any improvements in glycemic outcomes. Participants in the control group will use the Dexcom G6 CGM, the insulin dose capture system (Tempo pens and Tempo button), and the Data-logging Mode of DailyDose for the entire study. They will also be asked to complete a 30-minute aerobic exercise video at home once per week starting with the first 12-week period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of type 1 diabetes mellitus for at least 1 year.
2. Age 18 years and older.
3. Able to read, write and understand spoken English
4. HbA1c or GMI 7.5- 11.5% at screening. GMI (%) = 3.31 + 0.02392 × [mean glucose in mg/dL] based on prior 30 days of CGM data with at least 70% time CGM active[6]
5. Use of multiple daily insulin injections (MDI) for at least 30 days at the time of screening visit.
6. Willing to use the approved study insulin and devices while on study - Humalog and Basaglar Tempo pens, Dexcom G6 CGM, study iPhone, Apple watch
7. Willingness and ability to independently follow all study procedures, including attending all clinic and DSMES and behavioral health visits.
8. Total daily insulin requirements of less than 200 units

Exclusion Criteria:

1. Female of childbearing potential who is pregnant or intending to become pregnant or breast-feeding or is not using adequate contraceptive methods. Acceptable contraception includes birth control pill / patch / vaginal ring, Depo-Provera, Norplant, an IUD, the double barrier method (the woman uses a diaphragm and spermicide, and the man uses a condom), or abstinence.
2. History of stroke, heart failure, myocardial infarction, angina pectoris, or coronary arterial bypass graft or angioplasty.
3. Renal insufficiency (GFR < 60 ml/min, using either MDRD** or CKD-EPI# equation as reported by the laboratory).
4. Liver failure, cirrhosis, or any other liver disease that compromises liver function as determined by the investigator.
5. History of severe hypoglycemia during the 3 months prior to screening or hypoglycemia unawareness as judged by the investigator. Participants will complete a hypoglycemia awareness questionnaire. Participants will be excluded for four or more R responses.
6. History of diabetes ketoacidosis during the 3 months prior to screening, as diagnosed on hospital admission or as judged by the investigator.
7. History of psychiatric admission during the 6 months prior to screening.
8. Adrenal insufficiency.
9. Any active infection.
10. Known or suspected abuse of alcohol, narcotics, or illicit drugs.
11. Uncontrolled seizure disorder.
12. Active foot ulceration.
13. Severe peripheral arterial disease characterized by ischemic rest pain or severe claudication.
14. Major surgical operation within 30 days prior to screening.
15. Use of an investigational drug within 30 days prior to screening.
16. Chronic usage of any immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
17. Bleeding disorder, treatment with warfarin, or platelet count below 50,000.
18. Allergy to Humalog or Basaglar insulin.
19. Current chronic administration of oral or parenteral corticosteroids.
20. Any life-threatening disease, including malignant neoplasms and medical history of malignant neoplasms within the 5 years prior to screening (except basal and squamous cell skin cancer).
21. Initiation or titration of any medication used to lower glucose other than insulin in the 6 weeks prior to screening (e.g. metformin or semaglutide). Participants will not be excluded if they are non-insulin glucose lowering medication at a stable dose with no plans for discontinuation or dose modification during the course of the study). A positive response to any of the questions from the Physical Activity Readiness Questionnaire (see Appendix A) with one exception: participant will not be excluded if taking a single blood pressure medication and blood pressure is controlled on the medication (blood pressure is less than 140/90 mmHg).
22. Any chest discomfort with physical activity, including pain or pressure, or other types of discomfort.
23. Gastroparesis.
24. On a very low carbohydrate diet (less than 50g per day)
25. Taking part in another diabetes or obesity-related treatment study.
26. Any clinically significant disease or disorder which, in the opinion of the Investigator, may jeopardize the participant's safety or compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-05-15 (Estimated); Study Completion 2027-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in hemoglobin A1c (HbA1c) from baseline to 24 weeks after randomization | Enrollment and 24 weeks after randomization
  Hemoglobin A1c will be processed by a central lab. Lower values generally indicate better glucose control.

SECONDARY OUTCOMES:
Change in hemoglobin A1c (HbA1c) from baseline to 36 weeks after randomization | Enrollment and 36 weeks after randomization.
  Hemoglobin A1c will be processed by a central lab.
Change in percent of time in range (70-180 mg/dL) from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in range (70-180 mg/dL) from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in tight range (70-140 mg/dL) from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in tight range (70-140 mg/dL) from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in low glucose range (<70 mg/dL) from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in low glucose range (<70 mg/dL) from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in very low glucose range (<54 mg/dL) from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in very low glucose range (<54 mg/dL) from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in high glucose range (>180 mg/dL) from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in high glucose range (>180 mg/dL) from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in extreme high glucose range (>250 mg/dL) from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in percent of time in extreme high glucose range (>250 mg/dL) from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. Percent of time in this range during the two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in mean blood glucose from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. The average of values collected during the two weeks before a study time point will be treated as representing mean glucose at that study time point.
Change in mean blood glucose from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. The average of values collected during the two weeks before a study time point will be treated as representing mean glucose at that study time point.
Change in coefficient of variation of blood glucose from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. The coefficient of variation (CV) of CGM values is calculated as SD / mean * 100, where SD = standard deviation. The two weeks before a study time point will be used to represent that study time point.
Change in coefficient of variation of blood glucose from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  Continuous Blood Glucose Monitor (CGM) values are recorded every 5 minutes. The coefficient of variation (CV) of CGM values is calculated as SD / mean * 100, where SD = standard deviation. The two weeks before a study time point will be used to represent that study time point.
Change in Low Blood Glucose Index (LBGI) from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  The Low Blood Glucose Index (LBGI) is designed to reflect the risk of hypoglycemia and increases with the extent and frequency of hypoglycemic excursions. It is calculated by first taking f(BG) = (ln(BG)^1.084 - 5.381) for each blood glucose (BG) reading, then calculating rl(BG) = 22.7 * f(BG)^2 if f(BG) ≤ 0 and rl(BG) = 0 otherwise, and finally, by taking the average of the calculated rl(BG) values over all of the glucose readings measured in mg/dL.
Change in Low Blood Glucose Index (LBGI) from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  The Low Blood Glucose Index (LBGI) is designed to reflect the risk of hypoglycemia and increases with the extent and frequency of hypoglycemic excursions. It is calculated by first taking f(BG) = (ln(BG)^1.084 - 5.381) for each blood glucose (BG) reading, then calculating rl(BG) = 22.7 * f(BG)^2 if f(BG) ≤ 0 and rl(BG) = 0 otherwise, and finally, by taking the average of the calculated rl(BG) values over all of the glucose readings measured in mg/dL.
Change in High Blood Glucose Index (HBGI) from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  The High Blood Glucose Index (HBGI) is designed to reflect the risk of hyperglycemia and increases with the extent and frequency of hyperglycemic excursions. It is calculated by first taking f(BG) = (ln(BG)^1.084 - 5.381) for each blood glucose (BG) reading, then calculating rh(BG) = 22.7 * f(BG)^2 if f(BG) > 0 and rh(BG) = 0 otherwise, and finally, by taking the average of the calculated rh(BG) values over all of the glucose readings measured in mg/dL.
Change in High Blood Glucose Index (HBGI) from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  The High Blood Glucose Index (HBGI) is designed to reflect the risk of hyperglycemia and increases with the extent and frequency of hyperglycemic excursions. It is calculated by first taking f(BG) = (ln(BG)^1.084 - 5.381) for each blood glucose (BG) reading, then calculating rh(BG) = 22.7 * f(BG)^2 if f(BG) > 0 and rh(BG) = 0 otherwise, and finally, by taking the average of the calculated rh(BG) values over all of the glucose readings measured in mg/dL.
Change in T1-DDAS Core Score from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  The Type 1 Diabetes Distress Assessment System (T1-DDAS) Core Score is the average of 8 items on a scale from 1 to 5, where 1 is low distress and 5 is high distress associated with having type 1 diabetes.
Change in T1-DDAS Core Score from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  The Type 1 Diabetes Distress Assessment System (T1-DDAS) Core Score is the average of 8 items on a scale from 1 to 5, where 1 is low distress and 5 is high distress associated with having type 1 diabetes.
Change in T1-DDAS Management Difficulties Source Score from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  The Type 1 Diabetes Distress Assessment System (T1-DDAS) Management Difficulties Source Score is the average of 3 items rated from 1 to 5, where 1 is low distress and 5 is high distress. A higher score reflects higher distress related to management of type 1 diabetes.
Change in T1-DDAS Management Difficulties Source Score from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  The Type 1 Diabetes Distress Assessment System (T1-DDAS) Management Difficulties Source Score is the average of 3 items rated from 1 to 5, where 1 is low distress and 5 is high distress. A higher score reflects higher distress related to management of type 1 diabetes.
Change in T1-DDAS Hypoglycemia Concerns Source Score from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  The Type 1 Diabetes Distress Assessment System (T1-DDAS) Hypoglycemia Concerns Source Score is the average of 2 items rated from 1 to 5, where 1 is low distress and 5 is high distress. A higher score reflects higher distress related to hypoglycemia.
Change in T1-DDAS Hypoglycemia Concerns Source Score from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  The Type 1 Diabetes Distress Assessment System (T1-DDAS) Hypoglycemia Concerns Source Score is the average of 2 items rated from 1 to 5, where 1 is low distress and 5 is high distress. A higher score reflects higher distress related to hypoglycemia.
Change in T1-DDAS Technology Challenges Source Score from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  The Type 1 Diabetes Distress Assessment System (T1-DDAS) Technology Challenges Source Score is the average of 3 items rated from 1 to 5, where 1 is low distress and 5 is high distress. A higher score reflects higher distress related to using devices to manage type 1 diabetes.
Change in T1-DDAS Technology Challenges Source Score from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  The Type 1 Diabetes Distress Assessment System (T1-DDAS) Technology Challenges Source Score is the average of 3 items rated from 1 to 5, where 1 is low distress and 5 is high distress. A higher score reflects higher distress related to using devices to manage type 1 diabetes.

OTHER OUTCOMES:
Change in mean number of low glucose events / week from baseline to 24 weeks after randomization | Week 24 after randomization compared with baseline
  A single low glucose event is defined to start when the CGM drops below 70 mg/dL for at least three measurements and ends when the CGM rises above 69 mg/dL for at least three measurements. The two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in mean number of low glucose events / week from baseline to 36 weeks after randomization | Week 36 after randomization compared with baseline
  A single low glucose event is defined to start when the CGM drops below 70 mg/dL for at least three measurements and ends when the CGM rises above 69 mg/dL for at least three measurements. The two weeks before a study time point will be treated as representing blood glucose control at that study time point.
Change in total daily dose of insulin (units) from baseline to 24 weeks | Week 24 after randomization compared with baseline
  Insulin use will be tracked using bluetooth-enabled insulin pens. The two weeks before a study time point will be treated as representing that study time point.
Change in total daily dose of insulin (units) from baseline to 36 weeks | Week 36 after randomization compared with baseline
  Insulin use will be tracked using bluetooth-enabled insulin pens. The two weeks before a study time point will be treated as representing that study time point.
Change in total daily dose of insulin per kilogram (units/kg) from baseline to 36 weeks | Week 36 after randomization compared with baseline
  Insulin use will be tracked using bluetooth-enabled insulin pens. The two weeks before a study time point will be treated as representing that study time point.
Change in body weight measured at 36 weeks after randomization | Week 36 after randomization compared with baseline
  Maintaining or losing weight, rather than gaining, would be considered a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Leah Wilson, MD, Principal Investigator — Oregon Health and Science University
Locations (6):
- United States (6):
  - University of California, San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Barbara Davis Center, Aurora, Colorado
  - Joslin Diabetes Center, Harvard School of Medicine, Boston, Massachusetts
  - Mount Sinai School of Medicine, New York, New York
  - Oregon Health & Science University , Portland, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No
IPD cannot be shared due to concerns about participant privacy and confidentiality.